CLINICAL TRIAL: NCT07092163
Title: Evaluation of the Clinical Performance of 18-month Hybrid CAD/CAM Onlay Restorations: A Retrospective Study
Brief Title: Clinical Performance of Hybrid Computer-aided Design/Computer-aided Manufacturing (CAD/CAM) Onlay Restorations
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-29
Record Dates: First submitted 2025-07-18; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Indirect Posterior Restorations
Keywords: onlay; CAD/CAM; Qraypen; FDI criteria; overlay

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Description Hybrid CAD/CAM Onlay Group: Patients who received indirect onlay restorations fabricated from hybrid CAD/CAM blocks (Grandio Blocs, VOCO) on maxillary or mandibular molars between January 2023 and June 2023. Restorations were evaluated at baseline (1-week) and after 18 months using FDI clinical criteria and QLF imaging.
  Interventions: Device: QLF Imaging (Qraypen C®); Procedure: Clinical evaluation

INTERVENTIONS:
Device: QLF Imaging (Qraypen C®) — Fluorescence-based assessment of restoration margins using Qraypen C® device to measure autofluorescence loss (ΔF) and red fluorescence (ΔR). Imaging was performed during routine 18-month follow-up to detect micro-leakage or marginal biofilm activity.
Procedure: Clinical evaluation — Restorations were evaluated both at baseline (1-week recall) and at 18-month follow-up using the FDI World Dental Federation Clinical Evaluation Criteria, which allow structured and sensitive assessment of indirect restorations across three domains: Functional properties (e.g., marginal adaptation, fracture, retention, occlusion), Biological properties (e.g., recurrent caries, hypersensitivity, pulp status), Esthetic properties (e.g., marginal discoloration, surface texture, shade matching). Each criterion was scored on a 5-point ordinal scale: 1 = Clinically excellent / very good, 2 = Good (minor corrections), 3 = Satisfactory (acceptable with no significant clinical impact), 4 = Unsatisfactory (repair required), 5 = Clinically poor (replacement required). Scores of 1-3 were considered clinically acceptable, while scores of 4 or 5 indicated restorative failure.

SUMMARY:
Background: Hybrid Computer-Aided Design/Computer-Aided Manufacturing (CAD/CAM) materials have gained popularity in restorative dentistry due to their esthetic properties and favorable mechanical characteristics. However, clinical data evaluating the mid-term performance of indirect hybrid onlay restorations and their correlation with non-invasive fluorescence-based diagnostic tools remain limited. Aim: This study aimed to assess the 18-month clinical performance of indirect hybrid CAD/CAM onlay restorations using the World Dental Federation (FDI) criteria and to examine the diagnostic utility of Quantitative Light-induced Fluorescence (QLF) imaging in evaluating marginal adaptation, discoloration, and secondary caries. Materials and Methods: Thirty patients (aged 18-53) with a total of 33 maxillary or mandibular molar teeth restored using Grandio Blocs (VOCO, Germany) were retrospectively included. Restorations were clinically evaluated at baseline and 18 months using the FDI criteria (esthetic, functional, biological domains) by two calibrated, blinded observers. Standardized photographs, periapical radiographs, and QLF images were analyzed. QLF imaging was performed with Qraypen C® to quantify fluorescence loss (ΔF) and red fluorescence (ΔR) at restoration margins. Statistical analysis was conducted to determine the correlation between FDI scores and fluorescence parameters. Comparisons between baseline and 18-month FDI scores were performed using the Wilcoxon signed-rank test. The correlation between FDI evaluation scores and fluorescence parameters was assessed using the Spearman's rank correlation coefficient.A p-value of <0.05 was considered statistically significant for all tests.

DETAILED DESCRIPTION:
This retrospective clinical study was conducted at the Department of Restorative Dentistry, Faculty of Dentistry, Marmara University (approval number 2025-29). Patients who had their maxillary or mandibular molars treated with indirect hybrid Computer-Aided Design/Computer-Aided Manufacturing (CAD/CAM) onlay restorations by a clinician between January 2023 and June 2023 were included. All procedures were performed in accordance with the Declaration of Helsinki, and patients had previously provided institutional informed consent during hospital registration. The signed consent permitted the use of intraoral and extraoral radiographic images, digital records, clinical photographs, and other diagnostic materials for educational and scientific research purposes. A total of 58 buccal/lingual surfaces of the restoration-tooth margins of 33 molar teeth restored with Grandio Blocs (VOCO, Cuxhaven, Germany) were included in the evaluation. All hybrid onlay restorations included in the study were prepared and cemented by a faculty member with nine years of clinical experience in the Department of Restorative Dentistry. The eligibility of each tooth for onlay restoration was determined based on both clinical and radiographic evaluations. The criteria considered included the quantity and quality of the remaining tooth structure, occlusal relationships, periodontal status, history of pulpal or endodontic treatment, and esthetic demands. Tooth preparations were performed in accordance with standard adhesive protocols for hybrid onlays. A minimum of 2.0 mm occlusal reduction was ensured on both functional and non-functional cusps. Preparations featured a modified shoulder finish line, rounded internal line angles, and a convergence angle of approximately 10-15°, without any bevels. Prior to cavity preparation, the tooth shade was selected using the Vita Classical Shade Guide (VITA North America). Intraoral impressions were obtained with the Cerec Omnicam scanner (Dentsply Sirona), and the restorations were milled from Grandio blocs (VOCO) using a chairside CAD/CAM milling unit (CEREC MC X, Dentsply Sirona). The cementation procedure was performed in the same appointment as the cavity preparation and milling. Isolation was achieved using rubber dam, retraction cords, or cotton rolls as appropriate. The internal surface of the onlay was prepared with air abrasion using aluminum-oxide (Al2O3 particles, 53 μm particle size, 15 mm distance, 2.5 bar, 10 s; Velopex, London, UK), cleaned, dried, and silanized for 60 seconds. The prepared tooth surface was etched with 35% phosphoric acid, rinsed, and gently dried with air. Adhesive system (G-Premio Bond, GC Corp., Tokyo, Japan) was applied to both enamel and dentin surfaces and polymerized using light curing device (Demi Ultra, Kerr Dental, Orange, California, USA) for 20 s. The overlays were then bonded using a dual-curing resin cement (G-CEM One; GC Corp., Tokyo, Japan) in accordance with the manufacturer's instructions. Excess cement was removed with a dental scaler and floss. Light curing was performed for 20 s on each surface. Occlusal adjustments were completed using fine-grit diamond finishing burs under water cooling, followed by polishing with the Twist Diacomp Plus system (EVE Ernst Vetter GmbH, Birkenfeld, Germany). Patients were recalled one week later to reassess proximal contacts, marginal adaptation, and occlusal relationships. At the Department of Restorative Dentistry, follow-up controls for indirect hybrid CAD/CAM overlay restorations are routinely performed annually. During these visits, restorations are photographed using standardized protocols, and both periapical radiographs and fluorescence images are obtained. All image data are archived digitally for clinical monitoring and research purposes. Following the application of the inclusion and exclusion criteria, which encompassed the evaluation of clinical, radiographic and fluorescence values of 30 patients with 33 restorations between the ages of 18 and 53 were included in this study. All included restorations were evaluated at the baseline (1-week recall) and 18-month follow-up using the World Dental Federation (FDI) criteria (Hickel et al., 2010). Two blinded and calibrated observers (A.A.Ş and H.B.C) independently assessed the restorations across three primary domains (functional, biological, and esthetic). Each criterion was scored on a scale; 1 = clinically excellent/very good, 2 = good (after minor correction), 3 = clinically acceptable, 4 = clinically unsatisfactory (repair indicated), 5 = clinically poor (replacement required). Scores of 1-3 were considered clinically acceptable, whereas scores of 4 or 5 were interpreted as failures (Supplementary Table 1, 2 and 3). 18-month follow-up periapical radiographs were also analyzed. Prior to the assessments, observer calibration was performed. At the 18-month clinical recall, each restoration was assessed using Quantitative Light-induced Fluorescence (QLF) imaging acquired with the Qraypen C® device (AIOBIO, Seoul, South Korea), a fluorescence-based diagnostic tool with a field of view of 5-45 mm and a resolution of 1280 × 720 pixels. All images were obtained by a single calibrated operator (H.B.C) in a controlled clinical environment, where ambient lighting was minimized to ensure standardization across sessions. For each image, a region of interest (ROI) was manually defined around the tooth-restoration interface to allow consistent quantitative analysis. In line with the manufacturer's guidelines, the fluorescence assessment region was delineated to include only areas bordered by visually sound enamel and restoration. The fluorescence intensity within the ROI was evaluated using the manufacturer's proprietary software (QA2, version 1.24/1.25, Inspektor Research Systems BV, Amsterdam, The Netherlands). The key fluorescence parameters were measured: Autofluorescence loss (ΔFmax and ΔFaverage (%)), and red fluorescence (ΔRmax and ΔRaverage (%)). Statistical analysis was performed using IBM Statistical Package for the Social Sciences (SPSS) Statistics software. Descriptive statistics were calculated for all clinical and fluorescence parameters, including means, standard deviations, medians, and interquartile ranges, where appropriate. The normality of data distribution was assessed using the Shapiro-Wilk test. Comparisons between baseline and 18-month FDI scores were performed using the Wilcoxon signed-rank test for paired ordinal data. The correlation between FDI evaluation scores (marginal adaptation, marginal discoloration, and recurrent caries) and fluorescence parameters (ΔFmax, ΔFaverage, ΔRmax, ΔRaverage) was assessed using the Spearman's rank correlation coefficient. A p-value of <0.05 was considered statistically significant for all tests. Inter-examiner agreement for FDI scoring was evaluated using Cohen's kappa coefficient, with values greater than 0.85 considered indicative of high reliability.

ELIGIBILITY:
Inclusion Criteria:

* Received a single indirect onlay restoration fabricated from hybrid CAD/CAM material (Grandio Blocs)
* Restoration placed between January and June 2023 by a faculty member under standardized protocol
* Available 18-month clinical and fluorescence follow-up data (photos, radiographs, QLF)
* Signed institutional informed consent for use of medical records in research
* Adequate oral hygiene and regular dental attendance

Exclusion Criteria:

* Parafunctional habits (e.g., bruxism)
* Teeth with mobility (grade ≥1), active periodontal disease, or endodontic complications
* Pregnant or lactating individuals during treatment or follow-up
* Patients with systemic diseases affecting oral health (e.g., uncontrolled diabetes, immunosuppression)
* Incomplete clinical records or absence of follow-up data
* Restoration margins not extending supragingivally on at least one surface

Ages: 18 Years to 53 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients who had their maxillary or mandibular molars treated with indirect hybrid CAD/CAM onlay restorations by a clinician between January 2023 and June 2023 at the Department of Restorative Dentistry, Faculty of Dentistry, Marmara University were included.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
FDI Clinical Evaluation Score for Marginal Adaptation | At 1 week (baseline) and 18 months post-restoration
  Assessment of the functional integrity of the tooth-restoration interface using the revised FDI criteria.
  Scoring was performed by two calibrated observers (1 to 5 scale), where scores 1-3 were considered clinically acceptable, and 4-5 as failures.
FDI Clinical Evaluation Score for Marginal Discoloration | At 1 week (baseline) and 18 months post-restoration
  Esthetic assessment of the marginal staining at the restoration interface using short air-drying and visual inspection.
  Evaluated using the FDI esthetic domain A2; scores interpreted in terms of clinical acceptability.
FDI Clinical Evaluation Score for Secondary Caries | At 1 week (baseline) and 18 months post-restoration
  Biological evaluation of caries presence at the restoration margin using the FDI biological domain B1.
  Criteria based on air-drying, tactile probing, and radiographic findings.
ΔFaverage and ΔFmax (Loss of Fluorescence) at Restoration Margins | At 18-month follow-up
  Autofluorescence loss measured in percentage (%) using Qraypen C® and QA2 software.
  Indicates potential enamel demineralization around the margins. ROI (region of interest) was manually standardized per tooth.
ΔRaverage and ΔRmax (Red Fluorescence) at Restoration Margins | At 18-month follow-up
  Percentage increase in red fluorescence due to bacterial porphyrins. Used to evaluate microbial activity and biofilm accumulation at the restoration margin.

SECONDARY OUTCOMES:
Relationship Between FDI Scores and Red fluorescence (ΔRaverage, percentage increase) | At 18-month follow-up
  Statistical analysis between clinical evaluation scores (marginal adaptation, staining, and caries) and Red fluorescence (ΔRaverage, percentage increase). Evaluation used to assess consistency between objective fluorescence data and subjective clinical scoring.
Observer Agreement in FDI Scoring | Before data analysis at 18-month evaluation
  Inter-examiner reliability assessed via Cohen's Kappa coefficient for each FDI domain.
  A κ value > 0.85 was considered excellent agreement.
Relationship Between FDI Scores and autofluorescence (ΔFaverage, percentage decrease) | At 18-month follow-up
  Statistical analysis between clinical evaluation scores (marginal adaptation, staining, and caries) and autofluorescence (ΔFaverage, percentage decrease). Evaluation used to assess consistency between objective fluorescence data and subjective clinical scoring.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
When the study is published, it will be shared.
Supporting Information: Study Protocol, CSR